CLINICAL TRIAL: NCT00520858
Title: Effects of Exercise Modality on Abdominal Obesity and Health Risk Factors in Older Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ross2002
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- C (No Intervention)
- RE (Active Comparator): Resistance Exercise
  Interventions: Other: Resistance Exercise (RE)
- AE (Active Comparator): Aerobic Exercise
  Interventions: Other: Aerobic Exercise (AE)
- RAE (Active Comparator): Resistance and Aerobic
  Interventions: Other: Resistance and Aerobic Exercise (RAE)

INTERVENTIONS:
Other: Resistance Exercise (RE)
  Arms: RE
Other: Aerobic Exercise (AE)
  Arms: AE
Other: Resistance and Aerobic Exercise (RAE)
  Arms: RAE

SUMMARY:
The prevalence of abdominal obesity in the elderly is increasing at alarming rates and thus, requires immediate attention. By comparison to younger adults, obesity reduction in the elderly presents a unique challenge and requires an innovative approach. We propose a novel approach to investigate the effects of different exercise types as independent treatment strategies for the reduction of obesity and related health risk factors in older men and women. We propose that exercise without caloric restriction will be associated with modest weight loss (3-5%), that in turn will be associated with significant reduction in abdominal obesity, insulin resistance, and a corresponding increase in skeletal muscle mass and function. We will determine the separate effects of resistance and aerobic exercise on these primary outcome variables, and, whether a treatment strategy that combines the two is optimal.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 65 and 80 years of age.
* Men and women are self-sufficient, sedentary, abdominally obese (BMI between 27 and 34.9 kg/m2; waist circumference greater than 88 cm in women and 102 cm in men), weight stable (± 2 kg) for 6 months prior to the beginning of the study, be non-smokers, and not diabetic.
* We will study elderly women who are not taking hormone replacement therapy to create a homogeneous population in whom the effect of exercise on the principal outcome variables can be evaluated with minimal confounding.

Exclusion Criteria:

* Smokers and diabetics.
* Women taking hormone replacement therapy.

Ages: 65 Years to 80 Years | Sex: All
Age Groups: Older Adult
Enrollment: 145 (Actual)
Dates: Start 2003-09

PRIMARY OUTCOMES:
Abdominal obesity | 6 months

SECONDARY OUTCOMES:
Insulin Resistance | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Davidson LE, Hudson R, Kilpatrick K, Kuk JL, McMillan K, Janiszewski PM, Lee S, Lam M, Ross R. Effects of exercise modality on insulin resistance and functional limitation in older adults: a randomized controlled trial. Arch Intern Med. 2009 Jan 26;169(2):122-31. doi: 10.1001/archinternmed.2008.558. PMID 19171808